CLINICAL TRIAL: NCT01301742
Title: Relative Bioavailability of Single Dose BI 10773 Co-administered With Multiple Doses of 600 mg Gemfibrozil Bid Compared to Single Dose Treatment of BI 10773 Alone in Healthy Volunteers - a Phase I, Open-label, Randomised, 2-way Crossover Trial
Brief Title: Relative Bioavailability of Single Dose Empagliflozin (BI 10773) When Co-administered With Multiple Doses of 600 mg Gemfibrozil Compared to Single Dose Treatment With Empagliflozin (BI 10773) When Given Alone in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.58; 2010-023152-85 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Gemfibrozil

ARMS (2):
- BI 10773 (Active Comparator): Subject to receive one single dose BI 10773
  Interventions: Drug: BI 10773; Drug: Gemfibrozil
- BI 10773 plus gemfibrozil (Experimental): Subject to receive one single dose BI 10773 plus 600 mg gemfibrozil bid for 5 days
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 — 1 tablet single dose BI 10773 in the morning
  Arms: BI 10773
Drug: Gemfibrozil — Gemfibrozil 600 mg bid for 5 days
  Arms: BI 10773
Drug: BI 10773 — 1 tablet single dose BI 10773 in the morning
  Arms: BI 10773 plus gemfibrozil

SUMMARY:
To investigate the relative bioavailability of BI 10773 following coadministration with 600 mg gemfibrozil bid dosed to steady-state in comparison to BI 10773 when given alone.

ELIGIBILITY:
Inclusion criteria:

- Healthy male and female subjects

Exclusion criteria:

- Any finding of the medical examination (including Blood Pressure, Pulse Rate and Electrocardiogram) deviating from normal and of clinical relevance

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.58.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Macha S, Koenen R, Sennewald R, Schone K, Hummel N, Riedmaier S, Woerle HJ, Salsali A, Broedl UC. Effect of gemfibrozil, rifampicin, or probenecid on the pharmacokinetics of the SGLT2 inhibitor empagliflozin in healthy volunteers. Clin Ther. 2014 Feb 1;36(2):280-90.e1. doi: 10.1016/j.clinthera.2014.01.003. Epub 2014 Feb 1. PMID 24491572

RESULTS

PARTICIPANT FLOW:
Groups:
- Empa First, Then Empa and Gemfibrozil: Empagliflozin 25mg (Empa) was given as a single dose on Day 1, followed by a washout period of at least 7 days, followed by Gemfibrozil 600mg given twice daily for 5 days starting on day -2 and empa given as a single dose on Day 1, with gemfibrozil under steady-state conditions.
- Empa and Gemfibrozil First, Then Empa: Gemfibrozil 600mg was given twice daily for 5 days starting on day -2 and empagliflozin 25mg (empa) was given as a single dose on Day 1, with gemfibrozil under steady-state conditions. This was followed by a washout period of at least 7 days, followed by Empa given as a single dose on Day 1.
Period: First Intervention
Arm/Group | Empa First, Then Empa and Gemfibrozil | Empa and Gemfibrozil First, Then Empa
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout Period of at Least 7 Days
Arm/Group | Empa First, Then Empa and Gemfibrozil | Empa and Gemfibrozil First, Then Empa
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Empa First, Then Empa and Gemfibrozil | Empa and Gemfibrozil First, Then Empa
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: The two treatments given in a randomised order were:
  * Empagliflozin 25mg (Empa) was given as a single dose on Day 1
  * Gemfibrozil 600mg was given twice daily for 5 days starting on day -2 and empa was given as a single dose on Day 1, with gemfibrozil under steady-state conditions.
  Between treatments there was a washout period of at least 7 days.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Total Empa: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the plasma concentration-time curve of the analyte from time 0 extrapolated to infinity.
  The standard deviation presented in the analysis is actually the intra-individual geometric standard deviation (gCV).
Time Frame: 0 minutes (min), 20 min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 23h, 36h, 47h, 71h after the first dose
Population: PK set: All subjects who had taken at least 1 dose of trial medication who provided at least 1 observation for at least 1 primary pharmacokinetic (PK) endpoint without an important protocol violation with respect to the PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa Alone: Empagliflozin (Empa) 25mg given as a single dose on Day 1.
- Empa and Gemfibrozil: Gemfibrozil 600mg was given twice daily for 5 days starting on day -2 and empagliflozin 25mg (empa) was given as a single dose on Day 1, with gemfibrozil under steady-state conditions.
Arm/Group | Empa Alone | Empa and Gemfibrozil
Number analyzed (Participants) | 18 | 18
nmol*h/L | 4708.33 (7.5) | 7462.74 (7.5)
Statistical Analysis 1: Comparison: Empa Alone vs Empa and Gemfibrozil; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa and gemfibrozil divided by empa alone; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 158.50, 90% CI 2-sided [151.77 to 165.53], Standard Deviation 7.5 — Standard deviation is actually the intra-individual geometric coefficient of variation (gCV)

2. Primary Outcome: Total Empa: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of total Empagliflozin (Empa) in plasma, per period.
  The standard deviation presented in the analysis is actually the intra-individual geometric standard deviation (gCV).
Time Frame: 0 minutes (min), 20min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 23h, 36h, 47h, 71h after the first dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Alone | Empa and Gemfibrozil
Number analyzed (Participants) | 18 | 18
nmol/L | 602.24 (13.8) | 692.59 (13.8)
Statistical Analysis 1: Comparison: Empa Alone vs Empa and Gemfibrozil; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa and gemfibrozil divided by empa alone; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 115.00, 90% CI 2-sided [106.15 to 124.59], Standard Deviation 13.8 — Standard deviation is actually the intra-individual gCV

3. Secondary Outcome: Total Empa: Area Under the Curve 0 to Time of Last Quantifiable Data Point (AUC0-tz)
Description: Area under the plasma concentration-time curve of the analyte from time 0 to the time of the last quantifiable data point.
  The standard deviation presented in the analyses is actually the intra-individual geometric standard deviation (gCV).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Alone | Empa and Gemfibrozil
Number analyzed (Participants) | 18 | 18
nmol*h/L | 4643.81 (7.7) | 7350.84 (7.7)
Statistical Analysis 1: Comparison: Empa Alone vs Empa and Gemfibrozil; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa and gemfibrozil divided by empa alone; ANOVA; Based on ANOVA with terms for sequence, subjects within sequence, period and treatment; Geometric Mean Ratio = 158.29, 90% CI 2-sided [151.41 to 165.49], Standard Deviation 7.7 — Standard deviation is actually the intra-individual gCV

ADVERSE EVENTS:
Time Frame: First administration of trial medication until next administration of trial medication or up to post-study visit, 20 days
Groups:
- Gemfibrozil Alone: Between the first gemfibrozil administration and the empagliflozin administration, for the Empa and gemfibrozil treatment period.
Arm/Group | Empa Alone | Empa and Gemfibrozil | Gemfibrozil Alone
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 8/18 | 3/18 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa Alone (N=18) | Empa and Gemfibrozil (N=18) | Gemfibrozil Alone (N=18)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 4 | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes